CLINICAL TRIAL: NCT02829866
Title: THP AMIStem-H: Open, Retrospective and Prospective, Monocentric, Non Randomised Observational Study
Brief Title: AMIStem-H Radiographic Analysis
Status: Completed | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.001.11
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasty; Replacement; Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: AMIStem-H

SUMMARY:
Total hip replacement (THP) is widely used for hip osteoarthritis treatment. Surgeons are constantly looking to improve all aspects related to this procedure weather is improvement of implant design, instrumentation or surgical technique. Excellent clinical and radiological results were observed at medium and long term in the last years for AMIStem system.

This observational study has the objective to survey hip prosthesis stability and function of the operated hip in patients who are not exposed to surgical risks. The principal investigator will contact all patients in order to perform the follow-up visit according to standard practice. Patients operated between January 2010 and December 2011 will be invited in the study during the clinical visit organised according to standard practice. Preoperative clinical and radiological data, intraoperative details and postoperative follow-up data at 1-year will be retrospectively collected. Five-year and ten-year data will be prospectively collected after inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has received a total hip arthroplasty between January 2010 and December 2011
2. Patient who has received an AMIStem H femoral component
3. Patient who have signed the information letter in order to give agreement for the clinical data treatment

Exclusion Criteria:

1. Minor patient
2. Pregnant or breast feeding woman
3. Any patient who cannot or will not provide informed consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received a total hip arthroplasty with AMIStem H between January 2010 and December 2011 will be invited to participate in the study during the visit at 5 years previewed by standard practice.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Radiological analysis of radiolucency lines presence according to Gruen zone classification | 5 year

SECONDARY OUTCOMES:
radiological assessment of femoral deformation | 5 year, 10 year
radiological assessment of femoral stem subsidence | 5 year, 10 year
radiological assessment of cortical bone density | 5 year, 10 year
radiological assessment of calcar resorption | 5 year, 10 year
Radiological analysis of radiolucency lines presence according to Gruen zone classification | 10 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonspital Winthertur, Winterthur, Switzerland